CLINICAL TRIAL: NCT01670305
Title: Photodynamic Therapy and Periodontal Therapy. A Clinical, Microbiological and Immunoenzymatic Analysis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Marcio Zaffalon Casati, Professor, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0272.0.251.000-10
Record Dates: First submitted 2012-06-13; First posted 2012-08-22 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases | interventions — Photosensitizing Agents; Root Planing; Lasers; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Residual pocket - PDT (Experimental): Photosensitizer plus diiodo laser
  Interventions: Procedure: Residual pockets will be treated by laser + photosensitizer
- Residual pocket - Photosensitizer (Placebo Comparator): Photosensitizer alone
  Interventions: Procedure: Residual pockets will be treated only photosensitizer
- Residual pocket - SRP (Active Comparator): scaling and root planing alone
  Interventions: Procedure: Residual pockets will be treated scaling and root planing
- Furcation - PDT+SRP (Experimental): Photosensitizer plus diiodo laser associated with scaling and root planing
  Interventions: Procedure: laser + photosensitizer associated with scaling and root planing
- Furcation - SRP (Active Comparator): Photosensitizer associated with scaling and root planing
  Interventions: Procedure: furcation defects will be treated by scaling and root planing

INTERVENTIONS:
Procedure: Residual pockets will be treated by laser + photosensitizer — Experimental group: Residual pockets will be treated by laser + photosensitizer
  Arms: Residual pocket - PDT
Procedure: Residual pockets will be treated only photosensitizer — Placebo Comparator: Residual pockets will be treated only photosensitizer
  Arms: Residual pocket - Photosensitizer
Procedure: Residual pockets will be treated scaling and root planing — Active Comparator: Residual pockets will be treated scaling and root planing
  Arms: Residual pocket - SRP
Procedure: laser + photosensitizer associated with scaling and root planing — Experimental group: furcation defects will be treated by laser + photosensitizer associated with scaling and root planing
  Arms: Furcation - PDT+SRP
Procedure: furcation defects will be treated by scaling and root planing — Active Comparator: furcation defects will be treated by scaling and root planing
  Arms: Furcation - SRP

SUMMARY:
Residual pockets and furcation defects are challenging sites that require additional periodontal therapy. The aim of this study is evaluate 1)the effect of a single photodynamic therapy (PDT) as monotherapy residual pockets in single rooted teeth and 2) the effect of PDT in association with scaling and root planing (SRP) in class II furcation lesions with probing pocket depth (PPD) >5mm and bleeding on probing (BoP). A blind randomized controlled clinical trial was conducted in subjects presenting at least three residual pockets in single root teeth and subjects with at least one molar presenting class II furcation defect. To evaluate the effect of a single PDT as monotherapy in residual pockets, the selected sites were assigned to receive: PDT alone, photosensitizer alone or SRP alone. To evaluate the effect of PDT in association with SRP in class II furcation lesions, the selected sites were assigned to PDT+SRP or SRP alone. Clinical, microbiological and immunoenzymatic analyses were assessed at baseline, 3 and 6 months post-therapies.

DETAILED DESCRIPTION:
Residual pockets and class II furcation lesions are challenging sites that require additional periodontal therapy. The aims of this study were to evaluate:

1) the effect of a single PDT as monotherapy residual pockets in single rooted teeth and 2) the effect of PDT in association with SRP in class II furcation lesions.

A blind randomized controlled clinical trial was conducted in subjects presenting at least three residual pockets in single root teeth and subjects with at least one molar presenting class II furcation involvement.

To evaluate the effect of a single PDT as monotherapy in residual pockets, the selected sites were assigned to receive one of following therapies: PDT alone, photosensitizer alone or SRP alone.

To evaluate the effect of PDT in association with SRP in class II furcation lesions, the selected sites were assigned to receive PDT+SRP or SRP alone. Microbiological, immunoenzymatic analyses and clinical parameters: probing pocket depth (PPD), position of the gingival margin (PGM), relative clinical attachment level (RCAL), full mouth plaque (FMPS) and bleeding score (FMBS), will be assessed at baseline,3 and 6 months post-therapies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic periodontitis (according to the criteria of the 1999 international classification)
* at least three contralateral single rooted teeth with residual PPD > 5mm with bleeding on probing (BoP) in supportive periodontal therapy or with at least one molar presenting class II furcation defect.

Exclusion Criteria:

* pregnancy
* lactation
* current smoking and smoking within the past 10 years
* antibiotic therapies in the previous 6 months
* use of mouth rinses containing antimicrobials in the preceding 2 months
* systemic conditions that could affect the progression of periodontitis
* orthodontic appliances
* use of long-term administration of anti-inflammatory and immunosuppressive medications

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinical attachment level at 3 and 6 months. | baseline, 3 and 6 months post-therapies

SECONDARY OUTCOMES:
Probing Pocket depth | baseline, 3 and 6 months post-therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- School of dentistry - Paulista University UNIP, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www3.unip.br/default.asp